CLINICAL TRIAL: NCT06816589
Title: Using ChatGPT As a Job Coach for Adults with Autism Spectrum Disorder
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202307037RINA
Record Dates: First submitted 2025-02-04; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Autism; Job Interview Performance
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autism (Experimental)
  Interventions: Behavioral: ChatGPT-based job coaching

INTERVENTIONS:
Behavioral: ChatGPT-based job coaching — Using ChatGPT for creating job resumes, discussing job types, preparing and practicing for job interviews, writing job descriptions for individuals with Asperger's syndrome, and discussing workplace social interactions

SUMMARY:
The goal of this clinical trial is to examine the effectiveness of the ChatGPT-based job coach in helping ASD individuals prepare for job application, job interview, and interpersonal skills in workplaces. The main questions aim to answer are:

How can we develop a ChatGPT-based job coach system to assist individuals with autism spectrum disorder (ASD) in job applications, job interviews, and interpersonal skills in workplaces?

How effective is the ChatGPT-based job coach in helping ASD individuals (n=30) prepare for job applications, job interviews, and interpersonal skills in workplaces? What clinical correlates are associated with better effectiveness, and what are the interaction patterns between ASD adults and the ChatGPT platform?

Participants will complete assessment questionnaires (evaluating autism traits and empathy, approximately 30 minutes) and a one-hour job interview practice. Please follow the recommendations to use ChatGPT for completing your job resume, job type discussions, job interview preparation and practice, explanation of Asperger's traits for the workplace, and workplace social discussions. After one week of practice, you will fill out the assessment questionnaires and complete the job interview practice again.

ELIGIBILITY:
Inclusion Criteria:

* Young adult aged between 18 and 45 years who had a diagnosis of ASD from a licensed mental health or medical professional based on DSM-5;
* is motivated to have a job
* is able to use the ChatGPT on the computer under instruction (e.g., typing questions) and is able to provide feedback to the research team
* has a full-scale IQ > 70 on WAIS-IV
* scored ≧ 26 on the caregiver-reported Autism Spectrum Quotient (AQ), indicating clinical impairment associated with ASD
* agree to audio and video recording during the interview rehearsal.

Exclusion Criteria:

* A history of major psychiatric disorders (e.g., bipolar affective disorder, schizophrenia, or psychosis) or neurological diseases
* visual impairment and/or hearing impairment that would preclude participation in the study
* refuse audio and video recording during the interview rehearsal.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
the score of job interview role-play performance (JIRP) | 1 hour

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided